CLINICAL TRIAL: NCT02535728
Title: Anesthesia Geriatric Evaluation and the Prediction of Quality of Life in Elderly Cardiac Surgery Patients
Brief Title: Anesthesia Geriatric Evaluation and Quality of Life After Cardiac Surgery
Acronym: AGE
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, dr. P. Noordzij, dr. P. Noordzij, MD PhD, St. Antonius Hospital
Other Study IDs: NL53243.100.15
Record Dates: First submitted 2015-08-24; First posted 2015-08-31 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Quality of Life
Keywords: Frail Elderly; Cardiac Surgical Procedure; Risk Assessment; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples are taken directly after induction of anesthaesia.
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective observational cohort study to assess the predictive value of preoperative frailty on postoperative quality of life in cardiac surgery patients.

DETAILED DESCRIPTION:
Introduction:

The current population is ageing in a rapid pace. Currently elderly represent 17.8% of the Dutch population. Most recent estimates show this will increase to 25.6% 20 years' time. This rise in elderly will also reflect on the population of patients being referred for cardiac surgery. Especially elderly patients are at risk for postoperative complications, mortality or functional decline. In frail elderly this effect might be more pronounced. Frailty is an umbrella term that encompasses patient related factors such as weight loss, muscle wasting, inactivity, comorbidities and polypharmacy. Current scoring systems that are used to predict postoperative mortality and complications following cardiac surgery perform poorly in the elderly population and do not take into account frailty. Moreover they are designed to predict mortality and complications and are not validated to predict patient reported outcome measures such as quality of life or functional status. The aim of the AGE study is assess the value of frailty factors in predicting an improvement in quality of life one year after cardiac surgery.

Methods:

The AGE study is a prospective observational cohort study. All patients aged 70 years or older, scheduled for cardiac surgery, mentally competent and have signed informed consent are eligible for the study. During routine preoperative screening patients will be screened for frailty using different questionnaires and physical tests. The battery of tests exist of Short Form 36 (SF36), Multi Nutritional Assessment (MNA), Mini Mental State Examination (MMSE) and Nagi's scale for disability, Three physical tests: five meter walking speed, timed get up and go test and hand grip strength. A non-invasive measurement of Advanced Glycation Endproducts (AGEs) and a medication review. A blood sample will be taken to determine vitamin status, iron deficiency, pre-operative inflammatory parameters, CMV status, pneumococcal carriage and cardiac biomarkers. After surgery electronic patients charts will be studied to score postoperative complications or mortality. Three months and one year after cardiac surgery patients will receive SF-36 and World Health Organization Disability Assessment Schedule (WHODAS) 2.0 questionnaires to determine quality of life and functional status.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or older
* Mentally competent
* Planned cardiac surgery (coronary, valvular, rhythm, aortic or combination of those)
* Signed informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients planned for elective cardiac surgery and aged 70 years or older.
Sampling Method: Probability Sample
Enrollment: 577 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life Assessed by Short Form-36 (SF-36) | 12 months after surgery
  Assessed by Short Form-36 (SF-36)

SECONDARY OUTCOMES:
Quality of Life Assessed by Short Form-36 (SF-36) | 3 months after surgery
  Assessed by Short Form-36 (SF-36)
Psychosocial or physical functioning Assessed by World Health Organisation Disability Assessment Schedule 2.0 | 3 and 12 months after surgery
  Assessed by World Health Organisation Disability Assessment Schedule 2.0 (WHODAS 2.0)
Incidence of postoperative complications | 30 days after surgery
  Postoperative complications are scored according to Dutch national guidelines on reporting complications in cardiac surgery and include rethoracotomy, reoperation, bleeding, arrythmia, stroke, myocardial infarction, deep sternal wound infection, pneumonia, urinary tract infection, sepsis, respiratory insufficiency, prolonged respiratory support and renal failure (AKI).
Mortality | 30 days and 12 months after surgery
Length of stay in hospital and ICU | Post-Surgery. The expected length of stay in the ICU is 1 to 5 days and in hospital 5 to 10 days.
Postoperative delirium | 30 days
  Delirium according to intensive care delirium screening (ICDSC) or delirium observation screening (DOS)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Noordzij, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St Antonius hospital, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Background] Fruitman DS, MacDougall CE, Ross DB. Cardiac surgery in octogenarians: can elderly patients benefit? Quality of life after cardiac surgery. Ann Thorac Surg. 1999 Dec;68(6):2129-35. doi: 10.1016/s0003-4975(99)00818-8. PMID 10616989
- [Background] Chaturvedi RK, Blaise M, Verdon J, Iqbal S, Ergina P, Cecere R, deVarennes B, Lachapelle K. Cardiac surgery in octogenarians: long-term survival, functional status, living arrangements, and leisure activities. Ann Thorac Surg. 2010 Mar;89(3):805-10. doi: 10.1016/j.athoracsur.2009.12.002. PMID 20172133
- [Background] Ettema RG, Peelen LM, Kalkman CJ, Nierich AP, Moons KG, Schuurmans MJ. Predicting prolonged intensive care unit stays in older cardiac surgery patients: a validation study. Intensive Care Med. 2011 Sep;37(9):1480-7. doi: 10.1007/s00134-011-2314-1. Epub 2011 Jul 30. PMID 21805158
- [Background] Afilalo J, Mottillo S, Eisenberg MJ, Alexander KP, Noiseux N, Perrault LP, Morin JF, Langlois Y, Ohayon SM, Monette J, Boivin JF, Shahian DM, Bergman H. Addition of frailty and disability to cardiac surgery risk scores identifies elderly patients at high risk of mortality or major morbidity. Circ Cardiovasc Qual Outcomes. 2012 Mar 1;5(2):222-8. doi: 10.1161/CIRCOUTCOMES.111.963157. Epub 2012 Mar 6. PMID 22396586
- [Derived] Arends BC, Timmerman L, Vernooij LM, Verwijmeren L, Biesma DH, van Dongen EPA, Noordzij PG, van Oud-Alblas HJB. Preoperative frailty and chronic pain after cardiac surgery: a prospective observational study. BMC Anesthesiol. 2022 Jul 1;22(1):201. doi: 10.1186/s12871-022-01746-x. PMID 35778674
- [Derived] Verwijmeren L, Noordzij PG, Daeter EJ, Emmelot-Vonk MH, Vernooij LM, van Klei WA, van Dongen EPA. Preoperative frailty and one-year functional recovery in elderly cardiac surgery patients. J Thorac Cardiovasc Surg. 2023 Sep;166(3):870-878.e6. doi: 10.1016/j.jtcvs.2022.01.032. Epub 2022 Feb 3. PMID 35272845
- [Derived] Verwijmeren L, Bosma M, Vernooij LM, Linde EM, Dijkstra IM, Daeter EJ, Van Dongen EPA, Van Klei WA, Noordzij PG. Associations Between Preoperative Biomarkers and Cardiac Surgery-Associated Acute Kidney Injury in Elderly Patients: A Cohort Study. Anesth Analg. 2021 Sep 1;133(3):570-577. doi: 10.1213/ANE.0000000000005650. PMID 34153017
- [Derived] Verwijmeren L, Peelen LM, van Klei WA, Daeter EJ, van Dongen EPA, Noordzij PG. Anaesthesia geriatric evaluation to guide patient selection for preoperative multidisciplinary team care in cardiac surgery. Br J Anaesth. 2020 Apr;124(4):377-385. doi: 10.1016/j.bja.2019.12.042. Epub 2020 Feb 14. PMID 32063340